CLINICAL TRIAL: NCT01451814
Title: Development of Positive Psychotherapy for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor of Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-156241-1
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Smoking
Keywords: smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive psychotherapy (Experimental): 6 sessions of individual behavioral smoking cessation counseling that incorporates techniques from Positive Psychotherapy to increase positive affect and reduce negative affect prior to and after quitting smoking. Intervention includes 8 weeks of transdermal nicotine patch.
  Interventions: Behavioral: Positive Psychotherapy for smoking cessation; Drug: Nicotine polacrilex; Behavioral: Behavioral smoking cessation treatment
- Standard treatment (Active Comparator): 6 sessions of individual behavioral smoking cessation counseling with 8 weeks of transdermal nicotine patch. Inlcudes relaxation training to match time in the experimental condition
  Interventions: Drug: Nicotine polacrilex; Behavioral: Relaxation training; Behavioral: Behavioral smoking cessation treatment

INTERVENTIONS:
Behavioral: Positive Psychotherapy for smoking cessation — 6 sessions of individual behavioral smoking cessation counseling that incorporates techniques from Positive Psychotherapy to increase positive affect and reduce negative affect prior to and after quitting smoking. Intervention includes 8 weeks of transdermal nicotine patch.
  Arms: Positive psychotherapy
Drug: Nicotine polacrilex — 8 weeks of nicotine patch
Behavioral: Relaxation training — Instructions in progressive muscle relaxation
  Arms: Standard treatment
Behavioral: Behavioral smoking cessation treatment — Counseling on techniques to manage triggers and avoid smoking

SUMMARY:
The primary objective of this study is to test a manualized adaptation of positive psychotherapy (PPT) for smoking cessation (PPT-S). The investigators will conduct a preliminary randomized clinical trial (N = 80) to examine the feasibility, acceptability, and efficacy of PPT-S over 26 weeks of follow up in comparison to a standard smoking cessation treatment. Both treatments will be delivered in individual 6 sessions over 6 weeks, and will include provision of transdermal nicotine patch. The effect size estimates from this Stage 1b research will provide the foundation for a future application to conduct a large-scale, Stage II, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* smoke at least 5 cigarettes per day for longer than one year with no other ongoing tobacco product use
* willing to use the transdermal nicotine patch
* report at least a 5 on a 0 to 10 scale rating the importance of quitting smoking.

Exclusion Criteria:

* are currently experiencing psychotic symptoms, affective disorder (major depression, dysthymia, or mania) or substance use disorder (other than nicotine dependence)
* taking prescribed psychotropic medication or receiving other forms of psychotherapy
* concomitantly using other pharmacotherapies for smoking cessation
* have any contraindications for use of the transdermal nicotine patch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Result] Kahler CW, Spillane NS, Day AM, Cioe PA, Parks A, Leventhal AM, Brown RA. Positive Psychotherapy for Smoking Cessation: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2015 Nov;17(11):1385-92. doi: 10.1093/ntr/ntv011. Epub 2015 Feb 2. PMID 25646352

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Psychotherapy | Standard Treatment
Started | 35 | 31
Attended a Session | 35 | 31
Completed | 29 | 26
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Population: Participants fully eligible and attending the first session of counseling
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychotherapy | Standard Treatment | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (13.1) | 44.5 (13.8) | 46.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 35 | 29 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 29 | 25 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 66
Fagstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Score ranges from 0 to 10 with higher scores indicating greater dependence.
  units on a scale | 5.6 (2.4) | 5.4 (2.2) | 5.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 8 Weeks
Description: Biochemically verified abstinence from smoking over the past 7 days
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Positive Psychotherapy | Standard Treatment
Number analyzed (Participants) | 35 | 31
percentage of participants abstinent | 40.0 | 25.8
Statistical Analysis 1: Comparison: Positive Psychotherapy vs Standard Treatment; Test type: Superiority or Other; p = .22, Chi-squared; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.67 to 5.48]

2. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 16 Weeks
Description: Biochemically verified abstinence from smoking over the past 7 days
Time Frame: 16 Weeks
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Positive Psychotherapy | Standard Treatment
Number analyzed (Participants) | 35 | 31
percentage of participants abstinent | 22.9 | 6.5
Statistical Analysis 1: Comparison: Positive Psychotherapy vs Standard Treatment; Test type: Superiority or Other; p = .06, Chi-squared; Odds Ratio (OR) = 4.3, 95% CI 2-sided [0.84 to 22.1]

3. Primary Outcome: 7-day Point Prevalence Smoking Abstinence at 26 Weeks
Description: Biochemically verified abstinence from smoking over the past 7 days
Time Frame: 26 Weeks
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Positive Psychotherapy | Standard Treatment
Number analyzed (Participants) | 35 | 31
percentage of participants abstinent | 17.1 | 6.5
Statistical Analysis 1: Comparison: Positive Psychotherapy vs Standard Treatment; Test type: Superiority or Other; p = .18, Chi-squared; Odds Ratio (OR) = 3.0, 95% CI 2-sided [0.56 to 16.11]

ADVERSE EVENTS:
Arm/Group | Positive Psychotherapy | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychotherapy (N=35) | Standard Treatment (N=31)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No